CLINICAL TRIAL: NCT03974373
Title: Postoperative Evaluation of the Intraoral Technique of Buccal Fat Pad Removal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Metropolitana de Santos (Other)
Responsible Party: Principal Investigator, CAIO VINICIUS GONÇALVES ROMAN TORRES, Professor, Universidade Metropolitana de Santos
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SantosMU5
Record Dates: First submitted 2019-05-25; First posted 2019-06-04 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Bichat's Fat Pad Atrophy; Facial Expression
Keywords: Buccal mucosa
MeSH Terms: conditions — Facial Expression

STUDY DESIGN:
Intervention Model Description: We included in the present study 40 patients who sought the UNIMES Dentistry Clinic for the BFP removal procedure. All female, aged between 20 and 40 years and showing good general health. All the patients received information and had access to the informed consent form that after the necessary explanations was duly filled and signed.
  Clinical parameters such as periodontal indices (depth of probing, plaque index and gingival index), characteristics of the jugal mucosa, opening of the mouth, and the amount of fat removed were evaluated. After detailed anamnesis and verified the need to remove the fat ball by constant bite on the jugal mucosa or for aesthetic reasons of facial thinning the patients were instructed to perform the blood tests, fasting blood glucose and complete blood count. With the exams presenting normal levels and compatible with health status, the patients were scheduled to perform the proposed therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BFP removal (Experimental): this will be the group evaluated in this study, individuals who performed the BFP removal procedure.
  Interventions: Procedure: BFP removal

INTERVENTIONS:
Procedure: BFP removal — The surgical procedure was performed using the technique with intrabuccal access, already consecrated in the literature (Materasso 2006). The Bichat fat ball access was made by means of a small incision no more than 3 mm in length in the soft tissue located in the lower aspect of the zygomatic counterfoot, taking care to visualize and protect with the retractor the Stensen's conduit. With the aid of blunt-tipped or hemostatic scissors dissection was performed, taking care to preserve the membrane surrounding the ball of fat. After removal of one side, pressure was removed to remove air and the procedure was started on the opposite side, after the removal of the two sides was realized simple suture with silk thread. There were no formal indications for sending the samples for anatomic and / or histological examination.

SUMMARY:
In recent years there has been a growing number of procedures for the removal of the buccal fat pad (BFP) or as frequently referred to as bichectomy. Buccal fat pad removal can be used as part of the therapeutic procedure in cases of: sinus buco fistulas, peri-orbital defects, congenital palatal fissure, patients with severe bruxism, patients with constant lesions caused by bites on the jugal mucosa and in patients who are dissatisfied with the facial contour. In cases of thinning of the face, biting lesions and bruxism, total or partial of the BFP removal is performed, always taking into account a facial harmonization. The aim of the present study was to demonstrate the procedure of BFP removal and its respective postoperative period. A total of 40 BFP removal surgeries were performed between 2016 and 2017 with intraoral access technique. After the bichectomy procedure the subjects were followed for: 4, 7, 10, 15, 30, and 90 days. The postoperative period can be compared to that of a third molar extraction, and the use of analgesics and anti-inflammatories can adequately control the pain symptomatology. Edema and mouth opening limited for about 15 days were the most commonly found alterations in surgeries performed. The surgical technique is a simple and safe procedure provided by trained and experienced professionals. The bichectomy should be performed following a precise indication and the procedure is becoming a new area of practice for the dental surgeon, who can perform the procedure safely, reliably and with aesthetic and therapeutic results provided that with precise indications.

DETAILED DESCRIPTION:
The investigators included in the present study 40 patients who sought the UNIMES Dentistry Clinic for the BFP removal procedure. All female, aged between 20 and 40 years and showing good general health. All the patients received information and had access to the informed consent form that after the necessary explanations was duly filled and signed. Clinical parameters such as periodontal indices (depth of probing, plaque index and gingival index), characteristics of the jugal mucosa, opening of the mouth, and the amount of fat removed were evaluated. After detailed anamnesis and verified the need to remove the buccal fat pad by constant bite on the jugal mucosa or for aesthetic reasons of facial thinning the patients were instructed to perform the blood tests, fasting blood glucose and complete blood count. With the exams presenting normal levels and compatible with health status, the patients were scheduled to perform the proposed therapy. The surgical procedure was performed using the technique with intrabuccal access, already consecrated in the literature (Materasso, 2006). The buccal fat pad access was made by means of a small incision no more than 3 mm in length in the soft tissue located in the lower aspect of the zygomatic counterfoot, taking care to visualize and protect with the retractor the Stensen's conduit. With the aid of blunt-tipped or hemostatic scissors dissection was performed, taking care to preserve the membrane surrounding the ball of fat. After removal of one side, pressure was removed to remove air and the procedure was started on the opposite side, after the removal of the two sides was realized simple suture with silk thread. There were no formal indications for sending the samples for anatomic and / or histological examination. Patients were adequately medicated with analgesics and anti-inflammatories and antibiotics for 5 days. Kinesio therapy tapes were applied and placed towards the origin for insertion of the muscles involved in the region, and exchanged after 4, 7, and 10 days. Severe bilateral cryotherapy in the areas of extraoral surgery for 24 to 48 hours was performed. The first return was 4 days after the procedure and the next 7, 10, 15, 30, and ninety days, where physical, clinical, standardized photos and oral opening measurements were performed.

ELIGIBILITY:
Inclusion Criteria:

* patients with constant lesions caused by bites on the jugal mucosa
* patients who are dissatisfied with the facial contour.

Exclusion Criteria:

* any systemic problem
* altered blood tests
* presence of oral infection

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2019-05-05 (Actual)

PRIMARY OUTCOMES:
Limitation of mouth opening after the surgical procedure | 90 days
  to evaluate during the post-operative period the limitation of mouth opening, by means of manual pachymeter, and measured in millimeters.
presence of local edema | 90 days
  to evaluate in the post-operative period the presence of local edema. the presence of local edema will be verified through the patient's report, and the researcher's preservation through the photographs obtained in the preoperative period.
The facial contour was modified in the malar region after the surgical procedure. | 90 days
  photographs obtained before and after the surgical procedure will be placed in the PortraitPro 11 software and assessed for facial contour. The observed difference will be measured in millimeters

CONTACTS AND LOCATIONS:
Overall Officials: CAIO VINICIUS GONÇALVES R TORRES, Principal Investigator — Universidade Metropolitana de Santos
Locations (1):
- Caio Vinicius Gonçalves Roman Torres, Santos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
the study participants allowed the use of data only for this study and for this researcher

REFERENCES:
- [Background] Matarasso A. Managing the buccal fat pad. Aesthet Surg J. 2006 May-Jun;26(3):330-6. doi: 10.1016/j.asj.2006.03.009. PMID 19338917
- [Result] Matarasso A. Commentary on: Buccal Fat Pad Excision: Hydrodissection Technique. Aesthet Surg J. 2019 Sep 13;39(10):1046-1047. doi: 10.1093/asj/sjz086. No abstract available. PMID 31073600